CLINICAL TRIAL: NCT00596167
Title: Intradialytic Drug Removal by Short-daily Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0609-18
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: End Stage Renal Disease; Infection
Keywords: Short-daily hemodialysis; pharmacokinetics; levofloxacin; gentamicin; vancomycin
MeSH Terms: conditions — Kidney Failure, Chronic; Infections | interventions — Vancomycin; Levofloxacin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous antibiotics (Experimental): Intervention: administer intravenous vancomycin, gentamicin and levofloxacin. This study will determine the pharmacokinetics of intravenous vancomycin, gentamicin and levofloxacin in subjects receiving short-daily hemodialysis. There will not be a control arm for this study. The intervention for this arm will be to administer intravenous vancomycin, gentamicin and levofloxacin and draw blood samples at periodic intervals. The blood samples will be tested for these medications and pharmacokinetic analysis will be performed.
  Interventions: Drug: Intravenous antibiotics

INTERVENTIONS:
Drug: Intravenous antibiotics — Each subject will receive a single dose of 15 mg/kg vancomycin; 2 mg/kg gentamicin and 250 mg levofloxacin administered intravenously over a one-hour infusion period through the venous limb of their HD access (or tunneled catheter) via an IV pump.
  Other Names: Vancocin (vancomycin); Levaquin (levofloxacin); Gentamicin (gentamicin)

SUMMARY:
Short-daily hemodialysis is increasingly becoming a preferred alternative to the conventional intermittent (three times per week) hemodialysis schedule. Studies have shown that short-daily dialysis improves a patient's quality of life, high blood pressure, anemia and calcium-phosphorus balance. Infection, however, will likely remain a persistent problem for dialysis patients regardless of the frequency of treatments. There is currently a wealth of information to guide doctors on how much and how frequently to give an antibiotic for patients who receive intermittent (thrice weekly) hemodialysis. However, there is very little information on how to prescribe antibiotics for patient's receiving short-daily hemodialysis. This study will develop drug dose guidelines for patients receiving short-daily hemodialysis for three frequently used antibiotics, vancomycin, levofloxacin and gentamicin. These guidelines will assist doctors so that patients receive the most effective dose and frequency of an antibiotic to treat their infection.

The following is the study hypothesis which will be tested with two-sided, one sample t-tests comparing the AUC observed to historical measures8.

1) Vancomycin, levofloxacin and gentamicin are removed to a greater extent by short-daily hemodialysis than intermittent hemodialysis.

The following are the specific aims:

1. Determine the interdialytic pharmacokinetics of vancomycin, gentamicin, and levofloxacin by short-daily HD.
2. Determine the extent of vancomycin removal when administered during the last hour of short-daily HD.
3. Develop drug-dosing guidelines for vancomycin, gentamicin and levofloxacin for patients receiving short-daily HD.

DETAILED DESCRIPTION:
Despite improvements in dialysis machine and filter technology and refinements in providing an adequate "dose" of HD, patients receiving thrice-weekly hemodialysis (HD) have an alarming 20% annual mortality rate. Concomitant with this high mortality rate, patients with end stage renal disease (ESRD) also endure poorer qualities of life and medical complications such as anemia, infection, accelerated cardiovascular disease and bone disease associated with calcium-phosphorus disequilibrium. Recently, quotidian dialysis regimens, which include both the short-daily and nocturnal modalities, have emerged as dialytic approaches that appear to improve the patient's quality of life and attenuate the medical complications associated with ESRD1- 4. Specifically, recent studies have documented improvements in a patient's quality of life as measured by both general instruments (SF-36) and by renal disease specific tools. Short-daily HD regimens have also led to improvements in anemia allowing reductions in doses of erythropoietin. Similarly, in one study blood pressure control was improved with short-daily HD to such an extent that the majority of the study patients were eventually off of all antihypertensive medications. Phosphorus control has also improved with hemeral and especially nocturnal short-daily regimens. In one study of patients receiving nocturnal HD, all of the patients were completely weaned of their phosphorus binders and actually required intradialytic phosphorus supplementation. Finally, nutritional status also appears to be enhanced in studies of short-daily HD with increases in both appetite and weight gain observed. The medical benefits observed in these studies are believed to be secondary to the enhanced solute clearance and better extra-cellular volume management that short-daily HD affords as compared to intermittent HD. In particular, the nocturnal regimen appears especially effective since it provides a higher "dose" of HD than its hemeral counterpart.

According to the most recent United States Renal Data Service (USRDS) compilation, infection continues to exact a heavy toll among dialysis patients. The most recent USRDS mortality rate attributable to sepsis for dialysis patients was 27.0%. Despite the reported improvements in quality of life and medical complications provided by short-daily HD, infection will likely remain a persistent medical issue for dialysis patients. As a result, the appropriate provision of antibiotic therapy to patients receiving hemodialysis will remain paramount. Currently, there are no studies that have evaluated the pharmacokinetics of the commonly used antibiotics in the growing short-daily HD population. With no specific guidelines, pharmaco-kinetic estimations and frequent drug levels have been utilized to direct antibiotic dosing. This is likely not the best therapeutic approach and may not be the most cost-effective. This study will attempt to address this deficit in the clinical knowledge for three commonly used antibiotics, vancomycin, levofloxacin and gentamicin. The drug dosing guidelines developed from this study will ensure that this patient population receives the optimum antibiotic therapy to treat their infection in the most cost-effective manner.

Utilizing drug level data from an as yet unpublished study on the removal of gentamicin by thrice weekly dialysis, we configured the pharmacokinetic modeling software ADAPT to compare the serum levels of gentamicin during intermittent and short-daily HD. For the short-daily HD simulation, the ADAPT software demonstrated two periods of increased removal of gentamicin corresponding to the two sessions of short-daily HD (Figure 1). The purpose of the present study is to demonstrate in vivo that this is indeed true for gentamicin, as well as for vancomycin and levofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* currently receiving short-daily HD six times per week
* have no other acute intercurrent illness

Exclusion Criteria:

* history of a vancomycin, gentamicin or levofloxacin allergy
* weight within ± 30% of their ideal body weight
* Hgb < 10 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Decker, MD, PharmD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Decker BS, Kays MB, Chambers M, Kraus MA, Moe SM, Sowinski KM. Vancomycin pharmacokinetics and pharmacodynamics during short daily hemodialysis. Clin J Am Soc Nephrol. 2010 Nov;5(11):1981-7. doi: 10.2215/CJN.03450410. Epub 2010 Jul 8. PMID 20616157
- [Result] Decker BS, Mohamed AN, Chambers M, Kraus MA, Moe SM, Sowinski KM. Gentamicin pharmacokinetics and pharmacodynamics during short-daily hemodialysis. Am J Nephrol. 2012;36(2):144-50. doi: 10.1159/000339937. Epub 2012 Jul 18. PMID 22813936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Indiana University School of Medicine Short-daily hemodialysis clinic. The recruitment spanned 2007 to 2009. A total of six subjects were recruited.
Pre-assignment Details: Following completion of a subject's scheduled HD treatment, intravenous access will be maintained.
Groups:
- Intravenous Antibiotics: This study will have only one arm. This will be the experimental arm receiving the intravenous antibiotics, levofloxacin, vancomycin and gentamicin.
Period: Overall Study
Arm/Group | Intravenous Antibiotics
Started | 6 (All recruited subjects completed the study.)
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Antibiotics
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Intradialytic Clearance of Levofloxacin, Gentamicin and Vancomycin in Patients Receiving Short-daily Hemodialysis
Description: The intradialytic clearance of levofloxacin, gentamicin and vancomycin will be determined in patients receiving short-daily hemodialysis.
  (Of important note, due to technical issues the levofloxacin data was not able to be used for the analysis. Only the gentamicin and vancomycin data was analyzed.)
Time Frame: Serum concentrations for each drug will be determined from blood samples at 0 (pre-infusion), 30, 60 minutes (end of infusion).
Measure: Median (Full Range); unit: ml/min
Groups:
- Intravenous Antibiotic (Vancomycin): This study will have only one arm. All six participants in the study will receive an intravenous dose of the intravenous antibiotics, levofloxacin, vancomycin and gentamicin.
Arm/Group | Intravenous Antibiotic (Vancomycin)
Number analyzed (Participants) | 6
ml/min
  Intravenous antibiotic (vancomycin) | 7.2 [5.3 to 10]
  Intravenous antibiotic (gentamicin) | 7.6 [2.1 to 13.1]

ADVERSE EVENTS:
Time Frame: The incidence of adverse events was collected after the study drugs were infused and throughout the duration of the subjects' participation in the study (four days). After the subjects completed the study, there was no further monitoring.
Arm/Group | Intravenous Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Overall limitation is the relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes